CLINICAL TRIAL: NCT06348511
Title: XTics - A Gamified Enhancer of Non-Pharmacological Interventions in Tic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0165-22-TLV
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Tic Disorders
MeSH Terms: conditions — Tic Disorders

STUDY DESIGN:
Intervention Model Description: The study tested the impact of contingent and immediate reward (ICR) given by the game in respect to the participant's tic frequency relative to a random and non-contingent delayed reward (DR) provided by the end of the training day. Each participant underwent three training days in each of the the modes during one week. The training days included 3 (first day) or 4 (second and third days) game sessions. The order of the training modes was random.
Who Masked: Investigator
Masking Description: Personnel who interact directly with the study subjects were not aware of the assigned treatments. Personnel who analyze the data collected from the study are not aware of the treatment applied to any given group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate and contingent reward (ICR) (Experimental): Tic suppression directly affects gameplay, with participants informed that suppressing tics weakens opponents and improves card acquisition. Daily sessions end with feedback on suppression performance relative to that day's baseline.
  Interventions: Device: XTics
- Delayed reward (DR) (Active Comparator): The gameplay does not depend on performance, but participants still receive end-of-session feedback on tic suppression.
  Interventions: Device: XTics

INTERVENTIONS:
Device: XTics — XTics is a gamified protocol of behavioral treatment for tic disorders. The participant's tics are monitored in real-time and they are reflected as achievements in a game that the participant plays at the same time. The rewards aim to counteract processes that consolidate the tic. XTics is compatible with ERP treatment, and it includes an introductory psychoeducation session and three behavioral training sessions.

SUMMARY:
The investigators developed a neuroscientifically-informed gamified tic-therapy platform. The investigators previously identified tic-triggering elements in movies and video games. Next, the investigators employed these elements to generate and validate a gamified intervention protocol, which is based on a video game the investigators designed (called XTics). The study tests the efficacy of the gamified tool integrated in an exposure and response prevention (ERP) protocol to enhance both patient's compliance and clinical outcome.

DETAILED DESCRIPTION:
Background: Behavioral treatments are recommended as first-line interventions for tic disorders (TDs) in children and adults, which affect 2.99% of children. However, the effectiveness of these interventions is often undermined by the limited compliance especially of young individuals with the demanding treatment protocols. Addressing this issue, gamification of the treatment can enhance engagement and adherence in children. In the context of TDs, gamification provides significant additional benefits, particularly robust immediate feedback. This feedback can counteract the negative reinforcement processes, wherein the tic, believed to relieve the unpleasant premonitory urge, becomes consolidated. The investigators developed a gamified Protocol XTics, which leverages the previously untapped potential of combining various tic triggers with immediate reinforcement of tic suppression. The investigators evaluated the clinical value of XTics, focusing particularly on the benefits of immediate reward contingency in enhancing tic suppression performance.

Methods: The investigators developed a game incorporating tic triggers validated in a prior study. In one version of the game, its progression was influenced by real-time input from an experimenter who continuously monitored the participant's tics, rewarding tic suppression with favorable game outcomes. Employing a crossover design, the investigators trained 35 participants, aged 7-15, in both this version and another where the game's progression was independent of tic suppression. Following two online group Exposure and Response Prevention (ERP) training sessions, each participant engaged in three hourly sessions for each of the two conditions. Our evaluation focused on how the overall XTics protocol influenced tics and how this influence differed between the contingent and non-contingent versions of the game.

ELIGIBILITY:
Inclusion Criteria:

* Children and youths aged 7-15 years,
* At least moderate tic severity as indicated by a Yale Global Tic Severity Scale (YGTSS) tic severity score ≥ 11 and
* Tic frequency of over one tic per minute on average in the screening interview.

Exclusion Criteria:

* Behavioral treatment for tics in the past 12 months
* Pharmacological treatment for tics that has not been stable the for the past 6 weeks or with planned changes during study participation
* Evidence of tics that may produce physical harm to the child
* A history of psychiatric or neurological disorders requiring hospitalisation or a known cognitive decline.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The Tic Yale Global Tic Severity Scale (YGTSS) | Baseline (beginning of Week 1), after Phase 1 (beginning of Week 3), and after phase 2 (beginning of Week 5)
  A semi-structured clinical interview for assessment of tic severity administered to participants and parents. A clinician rates motor and vocal tics in terms of number, frequency, intensity, complexity and interference as well as overall related impairment over the preceding week. The investigators used YGTSS total tic severity scores.
The Parent Tic Questionnaire (PTQ) | Baseline, after Phase 1, after Phase 2, after the Booster phase (Week 7), and three months after the treatment termination
  A parent-report instrument for assessing tic severity. Tics are rated by frequency and intensity, and are summed to reflect motor, vocal, and total tics scores. PTQ has good internal consistency, good to excellent 2-week temporal stability, and convergent and discriminant validity in a clinic sample.
Premonitory Urge for Tic Scale (PUTS) | Baseline, after Phase 1, after Phase 2
  A self-report scale, which measures tic-related premonitory urges.
The Subjective Units of Distress Scale (SUDS) | By the end of each training day
  A self-reported questionnaire assessing the degree of inconvenience attributed to (1) tics and (2) the premonitory urges. Participants provided their ratings on a scale ranging from 0 (indicating absence) to 10 (indicating very severe). The total score was computed by summing the responses from both scales.
The "Urge Thermometer" | By the end of each training day
  A momentary ratings of the experienced magnitude of premonitory urge. The scale consisted of five qualitative descriptions of "0- not at all", "1 - weak", "2 - medium", "3 - strong" and "4- very strong". The child was instructed to pick a number/description to indicate his/her current pre-tic urge
Rush Videotape Protocol | Week 1, Week 3, Week 5
  Based on the Rush Videotape Protocol, the investigators recorded the participants under two resting epochs (i.e., performing no specific task) where they were left alone in the room and were instructed to remain seated and wait for 2.5 minutes while avoiding tic suppression. Tics were counted offline by a human rater who also marks epochs in which the participant is hidden or moved in a way that violated the instructions. The investigators used the total Rush scores, which combine scores for tic frequency (number of motor and phonic tics divided by duration of valid recording) and severity of motor and phonic tics.
Tic-to-tic interval | Week 1, Week 3
  The duration between two subsequent tics

SECONDARY OUTCOMES:
The Screen for Child Anxiety Related Emotional Disorders (SCARED) | Week 1, Week 5
  A self-report measure for screening anxiety disorders in children. Participants' ratings of their feelings over the previous two weeks are summed into scales of specific anxieties and general anxiety level. SCARED total score is used as a measure of anxiety symptoms. It was filled out by the child with the help of a parent.
The Children Depression Inventory (CDI) | Baseline and after Phase 2
  A commonly used self-report measure considered useful for screening comorbid depressive disorder in patients with TS (Snijders AH, Robertson MM, Orth M, 2006). The CDI total score is used as a measure of depression symptoms. It is filled out with the child. The investigators used five subscales: Negative Mood, Ineffectiveness, Anhedonia, Negative Self-Esteem, and Interpersonal Problems, as well as the global score.
The Conners' Parent Rating Scale-Revised Long Form (CRS:RL) | Week 1, Week 5
  The investigators used the long version, which contains 80 items and estimates different aspects of attention deficit and focus our analysis on the subscales of hyperactivity, inattention, and impulsivity and the composite of ADHD scores. It was filled out by parents or caregivers.
Obsessive Compulsive Inventory-Child Version (OCI-CV) | Week 1, Week 5
  OCI-CV estimates OCD severity across six domains of symptoms: Doubting/Checking, Obsessing, Hoarding, Washing, Ordering, Neutralizing. The total score was computed by summing the responses from all scales. It is filled out with the child. The investigatorslimited our analysis to Doubting/Checking, Obsessing, and total scores.
The Behavior Rating Inventory of Executive Function (BRIEF) | Week 1, Week 5
  BRIEF evaluates children's everyday executive functioning skills. Based on responses to 86 questions, executive functions are assessed across eight domains. The investigators used the composite Behavioral Regulation Index (BRI), which combines the Inhibit, Shift, and Emotional Control subdomains, the Metacognition Index (MI), which combines the subdomains of Organization of Materials and Monitor, and the overall Global Executive Composite (GEC) index, which combines the BRI and MI. BRIEF is filled out by the parents.
The Emotion Regulation Questionnaire (ERQ) | Week 1, Week 5
  A 10-item scale evaluating the respondents' tendency to regulate their emotions by cognitive Reappraisal or by expressive suppression. It was filled out by the child with the help of a parent.
User Engagement Scale (UES) | Week 3, Week 5
  The short Hebrew version of the UES is administered in regard to the game version they played in the past week. In this 12-item questionnaire, four different aspects of the user's experience are estimated using a five-point rating scale:(i) Focused attention, estimating the extent to which the user felt absorbed in the interaction and lost track of time; (ii) Perceived usability, indicating negative affect experienced as a result of the interaction and the degree of control and effort expended; (iii) Aesthetic appeal, i.e., the attractiveness and visual appeal of the interface; (iv) Reward factor, the extent to which the user felt that the experience was satisfying and interesting. The investigators used a composite index, which sums up the scores of UES scales.

CONTACTS AND LOCATIONS:
Overall Officials: Gal Raz, PhD, Principal Investigator — Sagol Brain Institute, Tel Aviv Sourasky Medical Center
Locations (1):
- Sagol Brain Institute, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No